CLINICAL TRIAL: NCT02659150
Title: A Multicenter, Open-Label, Proof-of-Activity Study of the Effect of Subcutaneous ACTEMRA on Inflamed Atherosclerotic Plaques in Patients With Rheumatoid Arthritis
Brief Title: Effect of Subcutaneous ACTEMRA on Inflamed Atherosclerotic Plaques in Patients With Rheumatoid Arthritis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated by sponsor owing to slow enrollment
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Ahmed Tawakol, Director, Nuclear Cardiology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML29520
Record Dates: First submitted 2015-12-21; First posted 2016-01-20 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Rheumatoid Arthritis
Keywords: tocilizumab; subcutaneous injection; rheumatoid arthritis; plaque inflammation; atherosclerotic plaque; joint inflammation; FDG-PET; PET-MR; ACTEMRA
MeSH Terms: conditions — Arthritis, Rheumatoid; Plaque, Atherosclerotic; Arthritis | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open-Label tocilizumab (Other): tocilizumab will be given to rheumatoid arthritis patients at a dose of 162 mg subcutaneously a week
  Interventions: Drug: tocilizumab

INTERVENTIONS:
Drug: tocilizumab — subjects will be treated with 162mg of weekly subcutaneous tocilizumab in an open-label manner, this will be done addition to MTX or monotherapy. On subsequent weeks after the first dose of tocilizumab, subjects will be instructed to inject the full amount of syringe according to the directions provided in the Instructions For Use (IFU).
  Other Names: ACTEMRA

SUMMARY:
The purpose of this study is to test the hypothesis that anti-IL-6 therapy is effective for reducing plaque inflammation as measured by fluorine-2-deoxy-D-glucose positron emission tomography (FDG-PET) in patients with rheumatoid arthritis (RA) who are synthetic disease-modifying antirheumatic drugs (dMARD) inadequate responders and are naive to biologic therapy.

DETAILED DESCRIPTION:
This multi-center study will recruit 21 subjects to undergo an open-label tocilizumab treatment for 13-18 weeks in order to examine the efficacy of tocilizumab on plaque inflammation in RA patients. This multi-center study will employ PET/MR imaging of the carotid and coronary arteries and aorta to assess the effect of anti-IL-6 therapy on arterial inflammation in patients with RA who are synthetic dMARD inadequate responders and are naive to biologic therapy.

Secondary, exploratory evaluation will also examine correlations between atherosclerotic plaque inflammation and the inflammatory activity of the rheumatoid joint measured by PET-MR imaging, as well as how the changes in inflammation correlate with lipid and inflammatory biomarkers, and how stress levels are associated with inflammatory activity.

Adults between 50 and 75 years old diagnosed with RA will come in for an initial screening visit to assess for clinical eligibility criteria (visit 1). During the screening period, patient acceptability for the study will be assessed on the basis of medical history, concomitant medications, physical examination, and clinical laboratory test results. The study doctor will review the screening test results and procedures to determine the subject eligibility prior to imaging. Women able to become pregnant will be excluded due to teratogenic side effects.

A FDG-PET/MR imaging study will be performed at a second screening visit (visit 2) to assess for the presence of arterial, plaque and joint inflammation. A serum pregnancy test will be drawn and confirmed to be negative prior to imaging for female subjects of childbearing potential. Acceptability for study participants will be confirmed on the basis of a tissue-to-background ratio (TBR) of greater than or equal to 1.7 in qualifying vessel (calculated using the mean of the maximum SUV) as measured from FDG-PET/MR imaging. Participants who meet clinical and imaging eligibility criteria will be enrolled into the study (visit 3). Subjects will receive first dose of tocilizumab subcutaneously, on subsequent weeks, subjects will be instructed to self-administer tocilizumab at a dose of 162mg every week for a 12 week period. 4 weeks post-initiation, participants will return for a clinical safety follow-up (visit 4). Final evaluation will include physical exams, clinical assessments and carotid IMT test. A second FDG-PET/MR imaging session will take place 12 weeks post-administration (visit 5).

Effect of tocilizumab on arterial plaque inflammation will be examined by measuring the change in FDG uptake in the carotid arteries, coronary arteries and aorta between the baseline and 12 week FDG-PET/MRI.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50-75
* Diagnosis of RA according to the revised 1987 American College of Rheumatology (ACR; formerly American Rheumatism Association), criteria.
* Patients who have had an inadequate response to non-biologic disease-modifying anti-rheumatic drug (DMARD) and are naïve to biologic agents.
* Presence of plaque inflammation, identified during secondary screening, defined as a target to baseline (TBR ratio) ≥ 1.7 in the carotid artery or ascending aorta.
* Not wheelchair or bedbound.
* At screening, active RA consisting of ≥4 swollen joints (28 joint count) and ≥ 4 tender joints (28 joint count) and any one of the following criteria:

  * Erythrocyte sedimentation rate (ESR) (Westergren) ≥ upper limit normal
  * CRP ≥ upper limit normal
* If using other non-biologic DMARDS, (ex: methotrexate, sulfasalazine, hydroxychloroquine, azathioprine, cyclosporine, leflunomide), patient must demonstrate inadequate response, be on stable dose(s) for at least 4 weeks prior to baseline visit. For methotrexate: patients must be on methotrexate for at least 3 months with 4 weeks stable dose, and will stay on stable dose during the study.
* taking corticosteroids, must be on stable doses of oral corticosteroids (≤ 10mg/day prednisone or equivalent) for at least 4 weeks prior to the baseline visit. Dose should remain stable throughout the study.
* Any investigational treatment not mentioned elsewhere must be discontinued for 4 weeks or 5 half lives, whichever is longer, prior to the baseline visit. Exposure to any investigational biologics should be discussed with the Sponsor.
* Signed informed consent (and informed assent of minor, if applicable).
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months after completion of treatment.
* Subject has provided written informed consent

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening.
* Previous treatment with any cell-depleting therapies, including investigational agents or approved therapies, some examples include: CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19 and anti-CD20.
* Treatment with intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of baseline.
* Immunization with a live/attenuated vaccine within 4 weeks prior to baseline.
* Previous treatment with TCZ or other biologics (an exception to this criterion may be granted for single dose exposure upon application to the PI on a case-by-case basis).
* Any previous treatment with alkylating agents such as chlorambucil, or with total lymphoid irradiation.
* Currently taking a statin
* An intra-articular injection of steroids within 6 weeks of imaging

Exclusions for General Safety:

* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies.
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease (including complicated diverticulitis, ulcerative colitis, Crohn's disease, or other symptomatic lower GI conditions that might predispose to perforations.)
* Diagnosis of liver disease or elevated hepatic enzymes, as defined by ALT, AST, or both > 1.5 x the upper limit of age-determined normal (ULN) or total bilirubin > ULN.
* Serum creatinine > 1.6 mg/dL (141 µmol/L) in female patients and > 1.9 mg/dL (168 µmol/L) in male patients. Patients with serum creatinine values exceeding limits may be eligible for the study if their estimated glomerular filtration rates (GFR) are >30
* Any history of recent serious bacterial, viral, fungal, mycobacterial or other opportunistic infections.
* Have serologic evidence of current or past HIV, Hepatitis B, or Hepatitis C.
* Positive QuantiFERON TB test , history of tuberculosis, or active TB infection without at least 4 weeks of adequate therapy for TB.
* Active infection with EBV as defined by EBV viral load ≥ 10,000 copies per mL of whole blood.
* Active infection with CMV as defined by CMV viral load ≥ 10,000 copies per mL of whole blood.
* Any of the following hematologic abnormalities, confirmed by repeat tests:
* White blood count <3,000/μL or >14,000/μL;
* Lymphocyte count <500/μL;
* Platelet count <100,000 /μL;
* Hemoglobin <8.0 g/dL; or
* Neutrophil count <2,000 cells/μL.
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
* Primary or secondary immunodeficiency (history of or currently active) unless related to primary disease under investigation.
* Any medical or psychological condition that in the opinion of the principal investigator would interfere with safe completion of the trial.
* History of other malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer.
* Pregnant women or nursing (breast feeding) mothers.
* Patients with reproductive potential not willing to use an effective method of contraception.
* History of alcohol, drug or chemical abuse within 1 year prior to screening.
* Neuropathies or other conditions that might interfere with pain evaluation unless related to primary disease under investigation.
* Rheumatic autoimmune disease other than RA, including SLE, MCTD, scleroderma, polymyositis, or significant systemic involvement secondary to RA (e.g., vasculitis, pulmonary fibrosis or Felty's Syndrome). Secondary Sjogrens syndrome with RA is allowable.
* Prior history of, or current inflammatory joint disease other than RA (e.g., gout, Lyme disease, seronegative spondyloarthropathy including reactive arthritis, psoriatic arthritis, arthropathy of inflammatory bowel disease).
* Relatively significant radiation exposure over the course of the year prior to randomization. Significant exposure is defined as:

  i) More than 2 PCI within 12 months of randomization ii) More than 2 myocardial perfusion studies within the past 12 months iii) More than 2 CT angiograms within the past 12 months iv) Any subjects with history of radiation therapy.
* Prior history of diverticulitis
* Contra-indications to MRI Imaging:
* Cardiac pacemaker that is not MRI compatible
* Surgical aneurysm clips
* Neurostimulator
* Implanted pumps
* Metal fragments in body / eyes
* Nitroglycerin patch that cannot be removed
* Colored contact lenses should not be worn in scanner
* Certain cochlear implants

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2019-11-16 (Actual); Study Completion 2019-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Tawakol, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Subject Enrollment
Arm/Group | Open-Label Tocilizumab
Started | 16
Completed | 11
Not Completed | 5
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 2
Period: Baseline Imaging
Arm/Group | Open-Label Tocilizumab
Started | 11
Completed | 9
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Period: Study Drug Dosing
Arm/Group | Open-Label Tocilizumab
Started | 9
Completed | 8
Not Completed | 1
Not completed — Adverse Event | 1
Period: Follow-up Imaging
Arm/Group | Open-Label Tocilizumab
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Screened and signed consent
Arm/Group | Open-Label Tocilizumab
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] — mean years (SD)
  years | 62.1 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Arterial Inflammation [Mean (Standard Deviation); unit: Target to Background Ratio (TBR)] — Population: 8 of 16 subjects completed imaging
  Target to Background Ratio (TBR)
    number analyzed (Participants) | 8
    (all) | 2.17 (0.56)

OUTCOME MEASURES:

1. Primary Outcome: Change in Arterial Inflammation in the Carotids
Description: The change in the target-to-background ratio of FDG uptake of the carotid, measured on PET-MR imaging before vs after 12 weeks of tocilizumab treatment. FDG uptake is calculated as Target to background values (TBR) . TBR, in turn, is calculated as the mean arterial standardized uptake value (SUV) divided by background blood pool SUV.
Time Frame: Baseline and 13-18 weeks follow-up
Population: subjects completing both imaging visits
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Open-Label Tocilizumab: tocilizumab was given to rheumatoid arthritis patients at a dose of 162 mg subcutaneously a week
  tocilizumab: subjects will be treated with 162mg of weekly subcutaneous tocilizumab in an open-label manner, this will be done addition to MTX or monotherapy. On subsequent weeks after the first dose of tocilizumab, subjects will be instructed to inject the full amount of syringe according to the directions provided in the Instructions For Use (IFU).
Arm/Group | Open-Label Tocilizumab
Number analyzed (Participants) | 8
Ratio | -0.10 (0.24)
Statistical Analysis 1: Comparison: Open-Label Tocilizumab; Paired T-test comparing values obtained during the follow-up imaging (at 13-18 weeks)minus the baseline values; Test type: Superiority; p = 0.26, t-test, 2 sided; Mean Difference (Final Values) = -0.10, Standard Deviation 0.24

2. Secondary Outcome: Association Between Change in Arterial Inflammation and Change in Articular Inflammation
Description: Change in FDG uptake in joints over the treatment period will be compared to the change in FDG uptake in arteries over the same period. FDG uptake is calculated as Target to background values (TBR)) . TBR, in turn, is calculated as the mean arterial standardized uptake value (SUV) divided by background blood pool SUV.
Time Frame: Baseline and 13-18 weeks follow-up
Population: participant who completed imaging
Measure: Number; unit: Correlation coefficient
Arm/Group | Open-Label Tocilizumab
Number analyzed (Participants) | 8
Correlation coefficient | 0.76
Statistical Analysis 1: Comparison: Open-Label Tocilizumab; correlation coefficient; Test type: Other; p = 0.036, Spearman; Spearman Correlation Coefficient = 0.76

3. Secondary Outcome: Change in Target to Background Ratio Within Carotid Artery Plaques
Description: Changes of Target to Background Ratio within the most diseased segment of the carotid arteries( a plaque-based analysis) before vs. after 12 weeks treatment
Time Frame: Baseline and 13-18 weeks follow-up
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Open-Label Tocilizumab
Number analyzed (Participants) | 8
Ratio | -0.58 (0.32)
Statistical Analysis 1: Comparison: Open-Label Tocilizumab; The carotid artery plaque with highest FDG uptake is located using Positron Emission Tomography/ Magnetic Resonance Imaging images. Thereafter Paired T- Test is used to compare baseline vs follow-up values of FDG uptake (before vs after 12 weeks of tocilizumab treatment). FDG uptake is assessed as a Target to background values (TBR) , which is calculated as the mean arterial standardized uptake value (SUV) divided by background blood pool SUV; Test type: Superiority; p = 0.14, t-test, 2 sided; Mean Difference (Final Values) = -0.19, Standard Deviation 0.32

4. Secondary Outcome: Association Between Change in Arterial Inflammation and Change in LDL
Description: Change in LDL over the treatment period will be compared to the change in FDG uptake in arteries over the same period. FDG uptake is calculated as Target to background values (TBR)) . TBR, in turn, is calculated as the mean arterial standardized uptake value (SUV) divided by background blood pool SUV.
Time Frame: Baseline and 13-18 weeks follow-up
Population: participant who completed imaging
Measure: Number; unit: Correlation coefficient
Arm/Group | Open-Label Tocilizumab
Number analyzed (Participants) | 8
Correlation coefficient | -0.66
Statistical Analysis 1: Comparison: Open-Label Tocilizumab; Test type: Superiority; p = 0.076, Spearman's Method; correlation coefficient = -0.66

5. Secondary Outcome: Association Between Change in Arterial Inflammation and Change in CRP
Description: Change in CRP (C-reactive protein) over the treatment period will be compared to the change in FDG uptake in arteries over the same period. FDG uptake is calculated as Target to background values (TBR)) . TBR, in turn, is calculated as the mean arterial standardized uptake value (SUV) divided by background blood pool SUV.
Time Frame: Baseline and 13-18 weeks follow-up
Population: participant who completed imaging
Measure: Number; unit: Correlation coefficient
Arm/Group | Open-Label Tocilizumab
Number analyzed (Participants) | 8
Correlation coefficient | 0.67
Statistical Analysis 1: Comparison: Open-Label Tocilizumab; Test type: Superiority; p = 0.07, Spearman's Method; Correlation coefficient = 0.67

6. Secondary Outcome: Correlation Between Change in BOLD Signals in the Amygdala and Anterior Cingulate Cortex With Atherosclerotic Plaque FDG Uptake
Description: Correlation coefficients cannot be calculated. The BOLD imaging was optional. Only one subject produced measurable BOLD imaging at baseline and follow-up. Thus while the data are analyzed, correlation coefficients cannot be calculated.
Time Frame: Baseline to 13-18 weeks follow-up
Population: Correlation coefficients cannot be calculated. The BOLD imaging was optional. Only one subject produced measurable BOLD imaging at baseline and follow-up. Thus while the data are analyzed, correlation coefficients cannot be calculated.
Measure: Number; unit: participants
Arm/Group | Open-Label Tocilizumab
Number analyzed (Participants) | 1
participants | NA — Correlation coefficients cannot be calculated. The BOLD imaging was optional. Only one subject produced measurable BOLD imaging at baseline and follow-up. Thus while the data are analyzed, correlation coefficients cannot be calculated for a single subject.

ADVERSE EVENTS:
Time Frame: 13-18 weeks
Arm/Group | Open-Label Tocilizumab
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 4/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Tocilizumab (N=16)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Tocilizumab (N=16)
elevated hepatic enzymes (Hepatobiliary disorders) | 1 (1) — Asymptomatic increase of AST and ALT to > 3x over normal without hyperbilirubinemia or jaundice. The abnormalities normalized rapidly after holding drug.
Leukopenia (Blood and lymphatic system disorders) | 1 (1) — minor transient reduction in blood counts.
Leukopenia and Throbocytopenia (Blood and lymphatic system disorders) | 1 (1) — minor reduction in PLT count
traumatic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — patient slipped on ice resulting in fracture
squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1) — recurrent squamous cell
Adenomiomatosys of the fundus of the gallbladder (Hepatobiliary disorders) | 1 (1) — Incidental finding on initial imaging prior to drug dosing
sinusitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Asymptomatic, incidental finding on imaging
cyst in the right kidney (Renal and urinary disorders) | 1 (1) — incidental finding on imaging
pericardial cyst (Cardiac disorders) | 1 (1) — incidental finding on imaging
vertebral hemangioma (Vascular disorders) | 1 (1) — incidental finding on imaging

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT02659150/Prot_SAP_000.pdf